CLINICAL TRIAL: NCT03730181
Title: Phase I/II Dose Finding and Safety Study of Rifapentine and Isoniazid in HIV-Infected and HIV-Uninfected Children With Latent Tuberculosis Infection
Brief Title: Tuberculosis Clinical Trials Consortium Study 35
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Stellenbosch (Other); Johns Hopkins University (Other); Sanofi (Industry); University of Cape Town (Other); Chris Hani Baragwanath Academic Hospital (Other); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6993
Record Dates: First submitted 2018-10-12; First posted 2018-11-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Latent Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis | interventions — rifapentine; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm Rifapentine and Isoniazid (Experimental): Single arm, open label and exposure-controlled. Intervention is rifapentine given in a new fixed dose combination once-weekly, in combination with isoniazid for 12 weeks, in HIV-infected and HIV-uninfected children aged 0-12 years in whom LTBI treatment is indicated. The protocol allows for parallel enrolment of children into cohorts 1 and 2, simultaneously, using a predetermined modeled initial dose for each cohort, separately. Similarly, cohorts 3 and 4 will be enrolled in parallel, using modeled doses for each cohort, based on data from cohorts 1 and 2 and historical data from TBTC trials.
  Interventions: Drug: Rifapentine; Drug: Isoniazid

INTERVENTIONS:
Drug: Rifapentine — Rifapentine. Initial dose will be 25mg/kg. Based on interim analysis, this may be adjusted throughout the study to achieve target exposures. The standalone water-dispersible rifapentine tablet may be used to adjust the rifapentine doses, if needed.
Drug: Isoniazid — Isoniazid. 25mg/kg

SUMMARY:
Hypotheses: Rifapentine (given as water-dispersible monolayer and/or fixed dose combination with isoniazid) dosing in HIV-infected and uninfected children ≤ 12 years of age with latent TB infection (LTBI) or with exposure to Mycobacterium tuberculosis (M. tuberculosis) will require higher mg/kg rifapentine dosing than adults to achieve adult- exposures which are correlated with efficacy in trials of TB prevention. Investigators further hypothesize that rifapentine will be safe and well-tolerated in HIV-infected and uninfected children who require treatment for LTBI.

DETAILED DESCRIPTION:
Design: Tuberculosis Trials Consortium Study 35 (TBTC S35) is a Phase I/II, open-label, single arm, exposure-controlled dose finding study using an adaptive design. S35 will evaluate the pharmacokinetics (PK), safety and tolerability of rifapentine given in a new fixed dose combination once-weekly, in combination with isoniazid for 12 weeks, in HIV-infected and HIV-uninfected children aged 0-12 years in whom LTBI treatment is indicated. The study utilizes a modified age de-escalation approach given the extensive PK and safety data already available in children older than 2 years of age. The protocol allows for parallel enrolment of children into cohorts 1 and 2, simultaneously, using a predetermined modeled initial dose for each cohort, separately. Similarly, cohorts 3 and 4 will be enrolled in parallel, using modeled doses for each cohort, based on data from cohorts 1 and 2 and historical data from TBTC trials.

Sample Size: Approximately 72 participants will be required to ensure a minimum number of 60 evaluable participants.

Participants will be enrolled in 4 age cohorts:

Cohort 1: ≥ 4 to ≤ 12 years Cohort 2: ≥ 24 months to < 4 years Cohort 3: ≥ 12 to < 24 months Cohort 4: 0 to <12 months

There will be a minimum of 12 participants each in cohorts 1 and 2, and 18 participants each in cohorts 3 and 4, to allow for 36 participants in the age group below 2 years, given the importance of developmental pharmacology in this youngest age group (Table 1) and the lack of historical data in this age group. Cohorts 3 and 4 will be enrolled once week 1 PK and safety data is available in cohorts 1 and 2.

Up to 18 HIV-infected children overall will be enrolled, with a target of 12 HIV-infected children overall. It is expected that most HIV-infected children will be > 3 years of age given current international recommendations regarding the use of efavirenz in children in international settings, where the study will be conducted. However, it is expected that integrase inhibitors (e.g. raltegravir) would become more routinely available during the study period, allowing younger HIV-infected children to also be enrolled on study.

Population: HIV-infected and uninfected children aged 0-12 years who could benefit from chemotherapy for LTBI to prevent the development of active tuberculosis, who have documented close recent exposure to a bacteriologically positive drug sensitive adult pulmonary TB source case, or who have proof of M. tuberculosis infection. HIV-infected children will be established on anti-retroviral therapy for at least 12 weeks prior to enrolment.

Sites:

TBTC Site 33, Desmond Tutu TB Centre, Department of Paediatrics and Child Health, Stellenbosch University, South Africa TBTC Site 34, Baragwaneth, Perinatal HIV Research Unit (PHRU), Wits Health Consortium, Soweto, Johannesburg, South Africa

Study Duration: Child participants will be on study for a total of 24 weeks, including a 12-week rifapentine and isoniazid dosing period, with an additional follow-up period of 12 weeks. The overall study accrual period will be approximately 18 months and the total study duration will be approximately 36 months.

Description of Agent or Intervention:

Participants will receive 12 once-weekly doses of water-dispersible rifapentine and isoniazid; the initial rifapentine dose in each age cohort will be determined based on historical population models and will be adjusted as data become available in paediatric cohorts in this study. Cohorts 1 and 2 will open up with a pre-selected modeled dose. Dose selection for cohorts 3 and 4 will be modeled from data emerging from cohorts 1 and 2 and historical data. Doses in cohorts will be adjusted as required based on interim PK and safety analyses. Isoniazid will be given at doses of up to 25 mg/kg, once weekly, in combination with pyridoxine (Vitamin B6) 25 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 0 - 12 years
2. Documented close (household or other close exposure) for at least an average 4 hours a day over the past 6 months to a bacteriologically confirmed adult (18 years or older) source case with pulmonary TB. The adult TB source case should have confirmed drug sensitive (sputum culture confirmed or XPERT MTB/Rif [Cepheid] positive TB and without any evidence of drug resistance, i.e., at least XPERT MTB/Rif rifampicin susceptible or an alternative molecular or phenotypic test indicating rifampicin susceptible M. tb) OR:
3. Evidence of M. tb infection (positive TST ≥ 10 mm in HIV-uninfected and TST ≥ 5 mm in HIV-infected participants or a positive commercial interferon-gamma release assay, as defined by the manufacturer)
4. Confirmed HIV status:

   HIV status will be confirmed by DNA PCR and Plasma HIV-RNA if the participant is <18 months of age.

   In participants ≥18 month of age HIV-ELISA testing will be completed. If any HIV test is positive in a child participant, regardless of age, the test result needs to be confirmed with a second HIV test, using HIV DNA or RNA PCR, from an independent sample.
5. HIV-infected participants should be on an ART regimen for at least 12 weeks prior to enrolment and should be clinically stable before entering the study, regardless of CD 4 count and HIV viral load. While on study, participants must be on an efavirenz- or raltegravir-based ART regimen which should have been given for at least 14 days prior to enrolment.
6. Caregiver (parent or legal guardian) gives written informed consent and assent from the child where applicable
7. Weight > 2.5 kg but < 40 kg

Exclusion Criteria:

1. Active TB disease (evidenced by: symptoms suggestive of TB, or suggestive findings on clinical examination, or suggestive chest radiographic findings, or positive mycobacterial culture/molecular TB tests -if culture/molecular testing was clinically indicated and was completed-, or currently on TB treatment for active disease).
2. Any documented drug resistant TB (DR TB) in an identified adult source case, defined as rifampicin resistance on Xpert or any other relevant approved molecular test, or phenotypic evidence of rifampicin resistance.
3. Receipt of a once-daily isoniazid regimen for > 30 days which was given for at least 14 consecutive days in the 30 days prior to enrolment.
4. Hb < 10 mg/dl
5. Weight for age z score below 2 or severe clinical malnutrition
6. Known allergy or hypersensitivity to isoniazid or rifapentine
7. Documented hepatic disorder including > 5 fold elevated upper limit of normal (ULN) ALT and/or bilirubin
8. Lansky play score < 50
9. Documentation of Hepatitis A or B infection
10. Female adolescents who have reached menarche will not be eligible.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Rifapentine exposure among participants by median area under the curve (AUC) | 12 weeks
  Target AUC is no more than 25% lower than, and no more than 75% higher than, the target AUC of 522 mcg*h/L. Data to be used for dose adjustments throughout the study and to create dosing algorithm for pediatric subgroups.

SECONDARY OUTCOMES:
Number of participants with Grade 3 or 4 adverse events | 24 weeks
  Cumulative number will be reported
Proportion of participants with Grade 3 or 4 adverse events | 24 weeks
  Cumulative proportion will be reported
Number of participants who discontinue study drug due to an adverse event | 12 weeks
  Cumulative number will be reported
Proportion of participants who discontinue study drug due to an adverse event | 12 weeks
  Cumulative proportion will be reported
Estimation of rifapentine absorption rate constant (ka) from plasma drug levels | 12 weeks
  Absorption rate constant will be estimated from plasma rifapentine blood levels, using population pharmacokinetic modeling methods. Models will be controlled for between-subject variability terms such as age and weight.
Estimation of rifapentine volume of distribution (Vd) from plasma drug levels | 12 weeks
  Volume of distribution will be estimated from plasma rifapentine blood levels, using population pharmacokinetic modeling methods. Models will be controlled for between-subject variability terms such as age and weight.
Estimation of rifapentine oral clearance (Cl/F) from plasma drug levels | 12 weeks
  Oral clearance will be estimated from plasma rifapentine blood levels, using population pharmacokinetic modeling methods. Models will be controlled for between-subject variability terms such as age and weight.
Post-hoc Bayesian prediction of rifapentine and metabolite peak concentration (Cmax) | 12 weeks
  Peak concentration will be predicted from plasma rifapentine and metabolite blood levels, using population pharmacokinetic modeling methods.
Post-hoc Bayesian prediction of rifapentine and metabolite time to peak concentration (Tmax) | 12 weeks
  Time to peak concentration will be predicted from plasma rifapentine and metabolite blood levels, using population pharmacokinetic modeling methods.
Post-hoc Bayesian prediction of rifapentine and metabolite area-under-the-curve (AUC0-24) | 12 weeks
  Area-under-the-curve will be predicted from plasma rifapentine and metabolite blood levels, using population pharmacokinetic modeling methods.
Post-hoc Bayesian prediction of rifapentine and metabolite half life (t 1/2) | 12 weeks
  Half life will be predicted from plasma rifapentine and metabolite blood levels, using population pharmacokinetic modeling methods.
Palatability scores | 12 weeks
  Using a standard validated Wong-Baker Faces tool which is a tool developed to help children communicate pain. For this outcome, the scale has been adapted to communicate like and dislike, and in-depth interviews
Acceptability scores | 12 weeks
  Using a standard validated Wong-Baker Faces tool which is a tool developed to help children communicate pain. For this outcome, the scale has been adapted to communicate like and dislike, and in-depth interviews
Incidence of tuberculosis | 24 weeks
  frequency of incident tuberculosis will be reported
Estimation of isoniazid absorption rate constant (ka) from plasma drug levels | 12 weeks
  Absorption rate constant will be estimated from plasma isoniazid blood levels, using population pharmacokinetic modeling methods. Models will be controlled for N-acetyltransferase 2 (NAT2) metabolizer genotype
Estimation of isoniazid volume of distribution (Vd) from plasma drug levels | 12 weeks
  Volume of distribution will be estimated from plasma isoniazid blood levels, using population pharmacokinetic modeling methods. Models will be controlled for N-acetyltransferase 2 (NAT2) metabolizer genotype
Estimation of isoniazid oral clearance (Cl/F) from plasma drug levels | 12 weeks
  Oral clearance will be estimated from plasma isoniazid blood levels, using population pharmacokinetic modeling methods. Models will be controlled for N-acetyltransferase 2 (NAT2) metabolizer genotype
Post-hoc Bayesian prediction of isoniazid peak concentration (Cmax) | 12 weeks
  Peak concentration will be predicted from plasma isoniazid blood levels, using population pharmacokinetic modeling methods, and accounting for N-acetyltransferase 2 (NAT2) metabolizer genotype
Post-hoc Bayesian prediction of isoniazid time to peak concentration (Tmax) | 12 weeks
  Time to peak concentration will be predicted from plasma isoniazid blood levels, using population pharmacokinetic modeling methods, and accounting for N-acetyltransferase 2 (NAT2) metabolizer genotype
Post-hoc Bayesian prediction of isoniazid area-under-the-curve (AUC0-24) | 12 weeks
  Area-under-the-curve will be predicted from plasma isoniazid blood levels, using population pharmacokinetic modeling methods, and accounting for N-acetyltransferase 2 (NAT2) metabolizer genotype
Post-hoc Bayesian prediction of isoniazid half life (t 1/2) | 12 weeks
  Half life will be predicted from plasma isoniazid blood levels, using population pharmacokinetic modeling methods, and accounting for N-acetyltransferase 2 (NAT2) metabolizer genotype

CONTACTS AND LOCATIONS:
Overall Officials: Anneke Hesseling, MD, Principal Investigator — University of Stellenbosch; Mark Cotton, MD, Principal Investigator — University of Stellenbosch; Avy Violari, MD, Principal Investigator — PHRU
Locations (1):
- Desmond Tutu TB Center, University of Stellenbosch, Stellenbosch, South Africa

REFERENCES:
- [Derived] Madzime RJ, van der Laan L, du Toit S, Barnabas S, Courtney I, Brown NE, Savic R, Solans BP, Dixon MG, Tsirizani L, Denti P, Boyd R, Hesseling AC; TBTC Study 35 team. Dolutegravir concentrations in children receiving 3-month weekly isoniazid and rifapentine (3HP) for tuberculosis prevention. Microbiol Spectr. 2026 Feb 3;14(2):e0330325. doi: 10.1128/spectrum.03303-25. Epub 2026 Jan 8. PMID 41504451